CLINICAL TRIAL: NCT06185933
Title: Lidocaine Spray vs Viscous Lidocaine Solution Plus Lidocaine Spray in Patients Undergoing Non-Sedated Esophagogastroduodenoscopy: A Randomized Controlled Trial
Brief Title: Lidocaine Spray vs Viscous Lidocaine Solution Plus Lidocaine Spray in Patients Undergoing Non-Sedated EGD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sawanpracharak hospital (Other)
Responsible Party: Principal Investigator, Natee Faknak, Clinical doctor at Department of medicine Sawanpracharak hospital, Sawanpracharak hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NF01
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pain; Satisfaction, Patient
Keywords: lidocaine spray; lidocaine solution; non-sedating EGD
MeSH Terms: conditions — Pain; Patient Satisfaction | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lidocaine spray alone (Active Comparator): patient in this arm will receive lidocaine spray five puffs of 10 % lidocaine spray (Xylocaine 10 % Spray, Astra Zeneca) (1 puff = 10 mg of lidocaine) 5 minutes before the start of the procedure
  Interventions: Drug: Lidocaine Spray
- receive lidocaine spray + lidocaine viscous solution (Active Comparator): patient in this arm will receive lidocaine spray + lidocaine viscous solution five puffs of 10 % lidocaine spray (Xylocaine 10 % Spray, Astra Zeneca) (1 puff = 10 mg of lidocaine) Plus 5 mL of 2 % viscous lidocaine solution (20 mg/mL) (Xylocaine 2 %, Astra Zeneca, London, UK)
  Interventions: Drug: Lidocaine Viscous+Lidocane spray

INTERVENTIONS:
Drug: Lidocaine Spray — Pharyngeal anesthesia using a topical lidocaine spray was administered in the preprocedure room, in the absence of the endoscopist or the research assistant. 5 minute before the UGE without any sedation
  Other Names: liocaine spray
  Arms: lidocaine spray alone
Drug: Lidocaine Viscous+Lidocane spray — Pharyngeal anesthesia using topical viscous lidocaine solution + lidocaine spray were administered in the preprocedure room, in the absence of the endoscopist or the research assistant. 5 minute before the UGE without any sedation
  Other Names: Lidocaine Viscous; Lidocane spray
  Arms: receive lidocaine spray + lidocaine viscous solution

SUMMARY:
This study aimed to compare the efficacy of lidocaine spray (S) alone versus lidocaine spray combined with lidocaine viscous solution (S+V) in facilitating pharyngeal observation during Non-sedating upper gastrointestinal endoscopy (UGE).

DETAILED DESCRIPTION:
A randomized controlled trial was conducted between July and October 2023 at Sawanpracharak hospital, Thailand. Of 250 patients undergoing UGE, 125 were randomly assigned to group S (lidocaine spray alone) and 125 to group S+V (lidocaine spray plus lidocaine viscous solution). The total dose of lidocaine did not exceed 5 mg/kg in both groups

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for upper gastrointestinal endoscopy:
* Patients who are robust, without chronic illnesses, or with controlled chronic conditions that do not adversely affect the function of any organ (American Society of Anesthesiologists (ASA) physical status classification I-II).

Exclusion Criteria:

* Has a history of receiving painkillers or sleeping pills within 24 hours before the endoscopy.
* Has a history of post-endoscopy nausea and vomiting.
* Patients who have undergone upper gastrointestinal endoscopy previously.
* Has chronic conditions such as epilepsy, vertigo, or mental health disorders.
* Has a history of allergy to anesthesia used in the study.
* Pregnant or currently breastfeeding.
* Refuses to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2024-07-04 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
procedural pain, measured using the visual analog scale (VAS). | 30 minute after finished precedure
  The procedural pain was evaluated using a visual analog scale (VAS, 0-10) with 0 being none and 10 being the most painfull

SECONDARY OUTCOMES:
patient tolerance | immediately after finished precedure
  1 = exceptional; 2 = well; 3 = fair; 4 = poor answer by endoscopist
endoscopist satisfaction | immediately after finished precedure
  1 = very satisfied; 2 = satisfied; 3 = neutral; and 4 = dissatisfied
patient satisfaction | 30 minute after finished precedure
  1 = very satisfied; 2 = satisfied; 3 = neutral; and 4 = dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Natee Faknak, Principal Investigator — Saawanpracharak hospital Thailand
Locations (1):
- Sawanpracharak hospital, Nakhon Sawan, Nakhonsawan, Thailand

IPD SHARING:
Plan to Share IPD: No